CLINICAL TRIAL: NCT06945666
Title: A Multicenter Prospective Study of Iguratimod in Combination With Tofacitinib in Patients With Rheumatoid Arthritis With Poor Response to Conventional or Biological DMARDs
Brief Title: A Study of Iguratimod in Combination With Tofacitinib in RA Patients
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Jie Chang (Other)
Responsible Party: Sponsor-Investigator, Jie Chang, Deputy Director, The Fourth Affiliated Hospital of Zhejiang University School of Medicine
Organization: The Fourth Affiliated Hospital of Zhejiang University School of Medicine (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KY-2025-072
Record Dates: First submitted 2025-04-02; First posted 2025-04-25 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2025-04

CONDITIONS: Rheumatoid Arthritis (RA
Keywords: iguratimod; tofacitinib
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — tofacitinib; Psychotherapy, Multiple; iguratimod

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- treatment group (Experimental): This study adopted a parallel controlled design, setting up a combined treatment group without an additional control group. The patients in the group received treatment with the standard dose of Iguratimod combined with tofacitinib. The recommended dose of Iguratimod is 25mg bid and that of tofacitinib is 5mg bid. During the treatment, other background therapeutic drugs were allowed to be used (determined by the prescribers), but other anti-rheumatic drugs that affected the study results were not allowed.
  Interventions: Drug: Combined therapy of Iguratimod and tofacitinib

INTERVENTIONS:
Drug: Combined therapy of Iguratimod and tofacitinib — This study aims to evaluate the efficacy and safety of the combination of iguratimod and tofacitinib in the treatment of RA patients with poor responses to traditional or biological DMARDs, providing evidence-based support for clinical treatment.
  Other Names: Combined therapy; Iguratimod and tofacitinib

SUMMARY:
Rheumatoid arthritis (RA) is a common chronic inflammatory autoimmune disease characterized by synovitis, which can cause joint pain, deformity, and extra-articular symptoms, seriously affecting the quality of life and lifespan of patients. Currently, the treatment of RA adopts a target attainment strategy, aiming to control the disease and reduce the disability rate. Although traditional disease-modifying antirheumatic drugs (DMARDs) can alleviate symptoms, they have slow onset, many side effects, and cannot completely stop the disease progression. Among biological DMARDs (bDMARDs), tumor necrosis factor-α (TNF-α) inhibitors have better effects, but some patients have poor responses and their conditions are not effectively controlled, thus new treatment options are urgently needed. This study aims to evaluate the efficacy and safety of the combination of iguratimod and tofacitinib in the treatment of RA patients with poor responses to traditional or biological DMARDs, providing evidence-based support for clinical treatment.

DETAILED DESCRIPTION:
This protocol is a multicenter, prospective study on the treatment of RA patients with poor response to conventional or biological DMARDs using a combination of iguratimod and tofacitinib. The study will be conducted simultaneously at 8 research centers, and each center will strictly follow the unified research protocol and standard operating procedures.

Researchers are not allowed to interfere with the treatment of patients. The treatment and follow-up arrangements are determined by the prescribing doctor based on the actual clinical situation. Enrolled patients receive standard-dose treatment with aramodine combined with tofacitinib. The recommended dose of iguratimod is 25mg twice a day, and the recommended dose of tofacitinib is 5mg twice a day. During the treatment period, other background treatment drugs (decided by the prescribing doctor) are allowed, but other anti-rheumatic drugs that may affect the research results are not allowed, in order to simulate the real clinical diagnosis and treatment environment to the greatest extent and ensure the extrapolation of the research results.

The observation period was from the time of patient enrollment to 24 weeks after the end of treatment. For patients who experienced serious adverse events (SAEs), follow-up was conducted until the outcome was clear or the study was terminated. During the study, the patients' disease conditions, adverse drug reactions, and other situations were closely monitored. At each follow-up visit, the researchers would record the patients' symptoms and signs in detail, conduct relevant laboratory tests and necessary imaging examinations, and comprehensively assess the patients' disease status and treatment effects.

This study adopts a parallel controlled design, setting up a combined treatment group without an additional control group. The focus is on evaluating the efficacy and safety of the combined treatment plan in the target patient population. Through multi-center collaboration, data from patients with different characteristics in various regions will be extensively collected to enhance the representativeness and reliability of the research results. Meanwhile, to ensure the quality of the research data, a complete data management and quality control system will be established. Regular audits and evaluations of the data from each center will be conducted to promptly identify and correct any issues in the data.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years old, male or female.
* Meets the classification criteria for rheumatoid arthritis established by the American College of Rheumatology (ACR) and the European League against Rheumatism (EULAR) in 2010.
* Meeting any of the following treatment conditions with poor efficacy (DAS28 score as moderate-high disease activity) : receiving conventional DMARDs therapy such as methotrexate for at least 3 months; Treatment with biological agents such as TNFi for at least 3 months; Treatment with eramode or tofaciib alone for at least 3 months.
* Understand the procedure and content of the test, and voluntarily sign the informed consent.

Exclusion Criteria:

* Patients with a known allergy to Iguratimod or tofacitinib.
* Patients who have previously used eramode or tofaciib and discontinued treatment for safety reasons;
* At the time of screening, they are in the acute phase of acute infection or chronic infection;
* At screening, hepatitis B DNA and/or hepatitis C RNA screening is positive, indicating viral hepatitis, HBs only Ag-positive healthy carriers were not considered as exclusion criteria, and inclusion of the patient was determined by the investigator;
* At the time of screening, have a history of active TB or TB screening suggests latent infection with mycobacterium tuberculosis;
* A medical condition or history of congestive heart failure at the time of screening;
* Include other ongoing projects or studies;
* Severe, progressive, uncontrolled disorders of vital organs and systems, as well as other medical conditions Any circumstances that should not be included in this collection.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2027-01-31 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
ACR20 (%) | 12 and 24 weeks of treatment
  American College of Rheumatology 20% improvement criteria (ACR20) response rates(Expressed as a percentage value) at 12 and 24 weeks of treatment.
ACR50 (%) | 12 and 24 weeks of treatment
  American College of Rheumatology 50% improvement criteria (ACR50) response rates(Expressed as a percentage value) at 12 and 24 weeks of treatment.
ACR70 (%) | 12 and 24 weeks of treatment
  American College of Rheumatology 70% improvement criteria (ACR70) response rates(Expressed as a percentage value) at 12 and 24 weeks of treatment.
DAS28 | 12 and 24 weeks of treatment
  Changes in disease activity score (DAS28) from baseline at 12 and 24 weeks of treatment. This score has no unit of measure.

SECONDARY OUTCOMES:
ESR (mm/h) | 4, 8, 12, and 24 weeks of treatment
  Changes in erythrocyte sedimentation rate (ESR, millimeters per hour) from baseline at 4, 8, 12, and 24 weeks of treatment.
CRP (mg/L) | 4, 8, 12, and 24 weeks of treatment
  Changes in C-reactive protein (CRP, milligrams per liter) levels from baseline at 4, 8, 12, and 24 weeks of treatment.
RF (IU/L) | 4, 8, 12, and 24 weeks of treatment
  Changes in rheumatoid factor (RF, international units per liter) levels from baseline at 4, 8, 12, and 24 weeks of treatment.
CCP (U/L) | 4, 8, 12, and 24 weeks of treatment
  Changes in anti-cyclic citrullinated peptide antibody (CCP, units per liter) levels from baseline at 4, 8, 12, and 24 weeks of treatment.
AE | From baseline to 24 weeks of treatment
  Incidence of adverse events (AE) of different severity

CONTACTS AND LOCATIONS:
Locations (1):
- 4th Affiliated Hospital, School of Medicine, Zhejiang University, Yiwu, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No